CLINICAL TRIAL: NCT01543750
Title: Phase 2 Study of 4-Aminopyridine for the Treatment of Episodic Ataxia Type 2
Brief Title: 4-Aminopyridine in Episodic Ataxia Type 2
Acronym: 4AP in EA2
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: University of Rochester (Other); University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CINCH-EA2; R01FD003923 (FDA)
Record Dates: First submitted 2011-05-27; First posted 2012-03-05 (Estimated); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Episodic Ataxia Type 2
Keywords: episodic ataxia; CACNA1A mutations
MeSH Terms: conditions — Episodic Ataxia, Type 2; Episodic Ataxia | interventions — 4-Aminopyridine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study Medication (Experimental): 4-aminopyridine 10mg twice daily for 8 weeks
  Interventions: Drug: 4-Aminopyridine
- Placebo (Experimental): placebo twice daily for 8 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 4-Aminopyridine
  Arms: Study Medication
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Episodic ataxia type 2 (EA2) is a rare familial neurological condition characterized by debilitating episodes of vertigo and imbalance. Since the serendipitous discovery of dramatic response of EA2 to acetazolamide, acetazolamide has been the first-line treatment for EA2. Yet, for those patients who do not respond to or cannot tolerate acetazolamide, there is no alternative treatment. The purpose of this randomized trial is to test whether 4-aminopyridine may reduce the ataxia episodes in EA2 as an alternative to acetazolamide. Funding Source - FDA OOPD

DETAILED DESCRIPTION:
This study aims to determine whether 4-aminopyridine (4AP) can reduce attacks of ataxia in patients with episodic ataxia type 2 (EA2), a rare but often debilitating condition. Episodic ataxia (EA) is a group of inherited disorders characterized by recurrent, discrete episodes of vertigo and ataxia variably associated with progressive ataxia. EA2, the most common and the best characterized of all the EA syndromes, is caused by heterozygous mutations in CACNA1A, which encodes the main subunit of a neuronal voltage-gated calcium channel, Cav2.1.

Although observational data suggest symptomatic resolution with acetazolamide in many EA2 patients, the investigators found in our patient databases that at least a third of the EA2 patients continue to suffer debilitating ataxia attacks, either because of incomplete control while on acetazolamide or because of intolerability or hypersensitivity to acetazolamide. For these patients there is no alternative intervention. 4-Aminopyridine (4AP) has been found to be helpful in a handful of patients with EA2. Recently, dalfampridine, an extended release formulation of 4AP (AMPYRA) by Acorda Therapeutics, received FDA approval to improve gait in multiple sclerosis.

The investigators plan to recruit 20 subjects with genetically defined EA2 who suffer frequent ataxia episodes (at least 3 episodes a month) to conduct a randomized trial of 4AP to examine its efficacy and tolerability in EA2. Study subjects will be recruited at UCLA and the University of Rochester to participate in a randomized, double-blind, double-crossover trial of 4AP.Each treatment period is 2-months with a 1-week wash-out period in between each treatment period. Participating subjects will undergo standardized history and physical examination at the time of enrollment. Participants will log their ataxia attacks daily by interactive voice response (IVR) system and will be interviewed monthly for events and side effects/toxicity. Study visits will occur at the beginning and the end of the study.

ELIGIBILITY:
Inclusion Criteria:

Patients will be included if they:

* Have EA2 genetically confirmed to harbor mutations in CACNA1A
* Are ≥ 18 years of age
* Are not taking acetazolamide (because of intolerance, poor response, or allergy)
* Are able to maintain a daily log of ataxia episode(s) and report daily by using an Interactive Voice Recording System (IVR) throughout the study
* Experience ≥ 3 ataxia episodes per month during the two-month screening period to qualify for randomization

Exclusion Criteria:

Patients will be excluded if they:

* Have seizures or a history of seizures
* Have first-degree relatives with EA2 and seizures
* Have renal disease with impaired function (Creatinine clearance CrCl≤50ml/min)
* Are pregnant or breast feeding (women of childbearing age will be tested for pregnancy and must be using birth control)
* Are unable to comply with the study requirement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
the frequency of ataxia episodes | 11 months
  Trial participants have frequent episodes of ataxia at baseline. The participants will document daily whether ataxia events occurred during the 2-month screening period and the 9-month study period by calling a toll-free number and participating in an Interactive Voice Response (IVR) system.

SECONDARY OUTCOMES:
impact on daily activities | 11 months
  Participants will use IVR to log the impact (on a scale of 0-3) of ataxia events, if any, on their daily activities:
  * (0) No impact
  * (1) Mild
  * (2) Moderate
  * (3) Severe
duration of ataxia episodes | 11 months
  Study Participants will use IVR daily to log the duration of ataxia events, if any, in hours.
severity of ataxia episodes | 11 months
  Study Participants will use IVR daily to log the severity of ataxia events, if any, on a scale of 1-9:
  (1) mild (9) very severe
treatment satisfaction | 9 months
  The study participant will respond by phone interview to the 11-item Treatment Satisfaction Questionnaire for Medication (TSQM Version 2) at the end of each of the four treatment periods.
Toxicity | 9 months
  The study participant will be interviewed by phone regarding toxicity using the [Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0] at two different time points (4 weeks, 8 weeks) of each 8-week Treatment Period. Spectrum and severity of toxicity and the prevalence among study participants will be documented.
Side Effects | 9 months
  The study participant will log side effects as they occur (reporting the seizures or other severe side effects immediately to Investigators) and will be interviewed by phone regarding side effects at two different time points (4 weeks, 8 weeks) of each 8-week Treatment Period. Spectrum of side effects and the prevalence among those treated will be documented.

CONTACTS AND LOCATIONS:
Overall Officials: Joanna C Jen, MD PhD, Principal Investigator — University of California, Los Angeles
Locations (3):
- United States (3):
  - University of California, Los Angeles (UCLA), Los Angeles, California
  - University of South Florida, Tampa, Florida
  - University of Rochester School of Medicine, Rochester, New York

REFERENCES:
- [Background] Atkinson MJ, Sinha A, Hass SL, Colman SS, Kumar RN, Brod M, Rowland CR. Validation of a general measure of treatment satisfaction, the Treatment Satisfaction Questionnaire for Medication (TSQM), using a national panel study of chronic disease. Health Qual Life Outcomes. 2004 Feb 26;2:12. doi: 10.1186/1477-7525-2-12. PMID 14987333
- [Background] Bever CT Jr, Young D, Anderson PA, Krumholz A, Conway K, Leslie J, Eddington N, Plaisance KI, Panitch HS, Dhib-Jalbut S, et al. The effects of 4-aminopyridine in multiple sclerosis patients: results of a randomized, placebo-controlled, double-blind, concentration-controlled, crossover trial. Neurology. 1994 Jun;44(6):1054-9. doi: 10.1212/wnl.44.6.1054. PMID 8208399
- [Background] DuMouchel W, Groer PG. A Bayesian methodology for scaling radiation studies from animals to man. Health Phys. 1989;57 Suppl 1:411-8. doi: 10.1097/00004032-198907001-00058. PMID 2606701
- [Background] Glasauer S, Strupp M, Kalla R, Buttner U, Brandt T. Effect of 4-aminopyridine on upbeat and downbeat nystagmus elucidates the mechanism of downbeat nystagmus. Ann N Y Acad Sci. 2005 Apr;1039:528-31. doi: 10.1196/annals.1325.060. PMID 15827015
- [Background] Griggs RC, Moxley RT 3rd, Lafrance RA, McQuillen J. Hereditary paroxysmal ataxia: response to acetazolamide. Neurology. 1978 Dec;28(12):1259-64. doi: 10.1212/wnl.28.12.1259. PMID 366453
- [Background] Imbrici P, Jaffe SL, Eunson LH, Davies NP, Herd C, Robertson R, Kullmann DM, Hanna MG. Dysfunction of the brain calcium channel CaV2.1 in absence epilepsy and episodic ataxia. Brain. 2004 Dec;127(Pt 12):2682-92. doi: 10.1093/brain/awh301. Epub 2004 Oct 13. PMID 15483044
- [Background] Harno H, Heikkinen S, Kaunisto MA, Kallela M, Hakkinen AM, Wessman M, Farkkila M, Lundbom N. Decreased cerebellar total creatine in episodic ataxia type 2: a 1H MRS study. Neurology. 2005 Feb 8;64(3):542-4. doi: 10.1212/01.WNL.0000150589.26350.3D. PMID 15699392
- [Background] Hoebeek FE, Stahl JS, van Alphen AM, Schonewille M, Luo C, Rutteman M, van den Maagdenberg AM, Molenaar PC, Goossens HH, Frens MA, De Zeeuw CI. Increased noise level of purkinje cell activities minimizes impact of their modulation during sensorimotor control. Neuron. 2005 Mar 24;45(6):953-65. doi: 10.1016/j.neuron.2005.02.012. PMID 15797555
- [Background] Jen J, Kim GW, Baloh RW. Clinical spectrum of episodic ataxia type 2. Neurology. 2004 Jan 13;62(1):17-22. doi: 10.1212/01.wnl.0000101675.61074.50. PMID 14718690
- [Background] Jen JC, Graves TD, Hess EJ, Hanna MG, Griggs RC, Baloh RW; CINCH investigators. Primary episodic ataxias: diagnosis, pathogenesis and treatment. Brain. 2007 Oct;130(Pt 10):2484-93. doi: 10.1093/brain/awm126. Epub 2007 Jun 15. PMID 17575281
- [Background] Jouvenceau A, Eunson LH, Spauschus A, Ramesh V, Zuberi SM, Kullmann DM, Hanna MG. Human epilepsy associated with dysfunction of the brain P/Q-type calcium channel. Lancet. 2001 Sep 8;358(9284):801-7. doi: 10.1016/S0140-6736(01)05971-2. PMID 11564488
- [Background] Lohle M, Schrempf W, Wolz M, Reichmann H, Storch A. Potassium channel blocker 4-aminopyridine is effective in interictal cerebellar symptoms in episodic ataxia type 2--a video case report. Mov Disord. 2008 Jul 15;23(9):1314-6. doi: 10.1002/mds.22071. PMID 18442126
- [Background] March B, Cardi T. Assessment of the cardiac safety of fampridine-SR sustained-release tablets in a thorough QT/QTc evaluation at therapeutic and supratherapeutic doses in healthy individuals. Expert Opin Investig Drugs. 2009 Dec;18(12):1807-15. doi: 10.1517/13543780903443096. PMID 19938897
- [Background] McEvoy KM, Windebank AJ, Daube JR, Low PA. 3,4-Diaminopyridine in the treatment of Lambert-Eaton myasthenic syndrome. N Engl J Med. 1989 Dec 7;321(23):1567-71. doi: 10.1056/NEJM198912073212303. PMID 2555713
- [Background] Ophoff RA, Terwindt GM, Vergouwe MN, van Eijk R, Oefner PJ, Hoffman SM, Lamerdin JE, Mohrenweiser HW, Bulman DE, Ferrari M, Haan J, Lindhout D, van Ommen GJ, Hofker MH, Ferrari MD, Frants RR. Familial hemiplegic migraine and episodic ataxia type-2 are caused by mutations in the Ca2+ channel gene CACNL1A4. Cell. 1996 Nov 1;87(3):543-52. doi: 10.1016/s0092-8674(00)81373-2. PMID 8898206
- [Background] Palermo TM, Valenzuela D, Stork PP. A randomized trial of electronic versus paper pain diaries in children: impact on compliance, accuracy, and acceptability. Pain. 2004 Feb;107(3):213-219. doi: 10.1016/j.pain.2003.10.005. PMID 14736583
- [Background] Sappey-Marinier D, Vighetto A, Peyron R, Broussolle E, Bonmartin A. Phosphorus and proton magnetic resonance spectroscopy in episodic ataxia type 2. Ann Neurol. 1999 Aug;46(2):256-9. doi: 10.1002/1531-8249(199908)46:23.0.co;2-6. PMID 10443893
- [Background] Smith W, Swan S, Marbury T, Henney H 3rd. Single-Dose pharmacokinetics of sustained-release fampridine (Fampridine-SR) in healthy volunteers and adults with renal impairment. J Clin Pharmacol. 2010 Feb;50(2):151-9. doi: 10.1177/0091270009344857. Epub 2009 Dec 4. PMID 19966074
- [Background] Spyker DA, Lynch C, Shabanowitz J, Sinn JA. Poisoning with 4-aminopyridine: report of three cases. Clin Toxicol. 1980 Jun;16(4):487-97. doi: 10.3109/15563658008989978. PMID 6250762
- [Background] Stefoski D, Davis FA, Faut M, Schauf CL. 4-Aminopyridine improves clinical signs in multiple sclerosis. Ann Neurol. 1987 Jan;21(1):71-7. doi: 10.1002/ana.410210113. PMID 2435223
- [Background] Stone AA, Shiffman S, Schwartz JE, Broderick JE, Hufford MR. Patient non-compliance with paper diaries. BMJ. 2002 May 18;324(7347):1193-4. doi: 10.1136/bmj.324.7347.1193. No abstract available. PMID 12016186
- [Background] Stone AA, Shiffman S, Schwartz JE, Broderick JE, Hufford MR. Patient compliance with paper and electronic diaries. Control Clin Trials. 2003 Apr;24(2):182-99. doi: 10.1016/s0197-2456(02)00320-3. PMID 12689739
- [Background] Strupp M, Schuler O, Krafczyk S, Jahn K, Schautzer F, Buttner U, Brandt T. Treatment of downbeat nystagmus with 3,4-diaminopyridine: a placebo-controlled study. Neurology. 2003 Jul 22;61(2):165-70. doi: 10.1212/01.wnl.0000078893.41040.56. PMID 12874393
- [Background] Strupp M, Kalla R, Dichgans M, Freilinger T, Glasauer S, Brandt T. Treatment of episodic ataxia type 2 with the potassium channel blocker 4-aminopyridine. Neurology. 2004 May 11;62(9):1623-5. doi: 10.1212/01.wnl.0000125691.74109.53. PMID 15136697
- [Background] van den Maagdenberg AM, Pietrobon D, Pizzorusso T, Kaja S, Broos LA, Cesetti T, van de Ven RC, Tottene A, van der Kaa J, Plomp JJ, Frants RR, Ferrari MD. A Cacna1a knockin migraine mouse model with increased susceptibility to cortical spreading depression. Neuron. 2004 Mar 4;41(5):701-10. doi: 10.1016/s0896-6273(04)00085-6. PMID 15003170
- [Background] van Diemen HA, Polman CH, van Dongen TM, van Loenen AC, Nauta JJ, Taphoorn MJ, van Walbeek HK, Koetsier JC. The effect of 4-aminopyridine on clinical signs in multiple sclerosis: a randomized, placebo-controlled, double-blind, cross-over study. Ann Neurol. 1992 Aug;32(2):123-30. doi: 10.1002/ana.410320203. PMID 1510353
- [Background] Vollmer T, Blight AR, Henney HR 3rd. Steady-state pharmacokinetics and tolerability of orally administered fampridine sustained-release 10-mg tablets in patients with multiple sclerosis: a 2-week, open-label, follow-up study. Clin Ther. 2009 Oct;31(10):2215-23. doi: 10.1016/j.clinthera.2009.10.007. PMID 19922892
- [Background] Vollmer T, Henney HR 3rd. Pharmacokinetics and tolerability of single escalating doses of fampridine sustained-release tablets in patients with multiple sclerosis: a Phase I-II, open-label trial. Clin Ther. 2009 Oct;31(10):2206-14. doi: 10.1016/j.clinthera.2009.10.008. PMID 19922891
- [Background] Walter JT, Alvina K, Womack MD, Chevez C, Khodakhah K. Decreases in the precision of Purkinje cell pacemaking cause cerebellar dysfunction and ataxia. Nat Neurosci. 2006 Mar;9(3):389-97. doi: 10.1038/nn1648. Epub 2006 Feb 12. PMID 16474392
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Weisz CJ, Raike RS, Soria-Jasso LE, Hess EJ. Potassium channel blockers inhibit the triggers of attacks in the calcium channel mouse mutant tottering. J Neurosci. 2005 Apr 20;25(16):4141-5. doi: 10.1523/JNEUROSCI.0098-05.2005. PMID 15843617